CLINICAL TRIAL: NCT05046470
Title: SARS-CoV-2 Transmission in Belgian Primary Schools of the Federation Wallonia - Brussels: An Epidemiological Pilot Study
Acronym: DYNAtracs
Status: Active, not recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: University of Liege (Other); Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/16NOV/552; ISRCTN16837012 (Registry Identifier: ISRCTN registry)
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: SARS-CoV-2 Infection
Keywords: Primary Schools
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators hypothesize that children are less likely to become infected in the school environment, compared to the household or outside the school setting. Primary schools do not play a major role in SARS-CoV-2 spreading. They hypothesize that incidence level in schools is mainly a consequence of community transmission. The incidence level in household and that the secondary attack rate in schools remains at least 5 times lower that the transmission level in households.

ELIGIBILITY:
Inclusion Criteria:

* All children and school attenders from selected schools was invited to participate

Exclusion Criteria:

* Refusal to provide written informed consent before enrolment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Belgian primary schools of the Federation Wallonia - Brussels that have organized a full resumption of school activities with the control measures recommended by the government, are eligible for the study.
  Twelve schools were chosen by purposive criteria: either high (≥2 classes per grade) or low size of the school, a school within an area with either a high or a low incidence of SARS-CoV-2 during April 2020, the first wave of covid-19 in Belgium, and a school with either a high or a low socioeconomic level (Belgian 20-point-scale ISE idex >14 or <6).
Sampling Method: Non-Probability Sample
Enrollment: 1233 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Infection of a child with SARS-CoV-2 secondary to a classmate | 6 weeks
  Time varying number and proportion of children infected with SARS-CoV-2 secondary to an asymptomatic infected classmate (transmission rate inside school with the child being the infector).
Infection of an adult school-attender with SARS-CoV-2 secondary to an infected child | 6 weeks
  Time varying number and proportion of adult school-attenders infected with SARS-CoV-2 secondary to an asymptomatic infected child (transmission rate inside school but from a child to an adult).
Infection of a child with SARS-CoV-2 secondary to an adult school attender | 6 weeks
  Time varying number and proportion of children infected with SARS-CoV-2 secondary to an infected adult school-attender (transmission rate inside school but from an adult to a child)
Infection of a child with SARS-CoV-2 secondary to a contact outside the school, including the household | 6 weeks
  Time varying number and proportion of children infected with SARS-CoV-2 secondary to a household contact or outside the school (transmission rate from in community).

CONTACTS AND LOCATIONS:
Overall Officials: Annie Robert, Pr, Study Director — Université Catholique de Louvain
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
All collected IPD

REFERENCES:
- See also: Protocol — https://www.sesa.ucl.ac.be/Dynatracs/assets/pdf/1011_ChildrenTransmission_Protocol_Ver1.0_10NOV20.pdf
- See also: Study website — https://www.sesa.ucl.ac.be/Dynatracs/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT05046470/Prot_SAP_000.pdf